CLINICAL TRIAL: NCT01608932
Title: RENEWING HEALTH - Telemonitoring of Elderly and Frail Patients With Multiple Chronic Diseases in Veneto Region
Brief Title: Life-long Monitoring of Frail Patients With Chronic Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regione Veneto (Other)
Collaborators: European Commission (Other); Local Health Authorities n. 4 (Unknown); Local Health Authorities n. 7 (Unknown); Local Health Authorities n. 9 (Unknown); Local Health Authorities n. 12 (Unknown); Local Health Authorities n. 13 (Unknown); Local Health Authorities n. 16 (Unknown); Local Health Authorities n. 20 (Unknown); SIMG (Italian College of General Medicine) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: G.A. 250487 - Veneto WP8Cl10
Record Dates: First submitted 2012-05-29; First posted 2012-05-31 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2012-05

CONDITIONS: Multiple Chronic Diseases Among Diabetes Mellitus, Chronic Obstructive Pulmonary Diseases and Heart Failure
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (No Intervention): Treatment as usual
- Telemonitoring for frail patients with chronic diseases (Experimental): Telemonitoring for frail patients with chronic diseases
  Interventions: Procedure: Telemonitoring for frail patients with chronic diseases

INTERVENTIONS:
Procedure: Telemonitoring for frail patients with chronic diseases — Patients are equipped with a telemonitoring kit that can be composed by a portable wrist clinic device, a digital weight scale and a glucometer for clinical parameters measuring, according to the pathologies of the patient. The equipment is completed by a gateway device for data transmission.
  The patient can monitor a complete set of clinical parameters, such as pulse-oxymetry, heart rate, blood pressure, ECG, body weight and glycemia with a frequency set by the clinician in the personalized treatment plan. In the same protocol the clinician includes also the alarm thresholds that determine when the clinical measures are out-of-range. Data are transmitted to a regional eHealth centre where a group of operators keeps these information under control and alerts the general practitioner in case of worsening of symptoms.
  Arms: Telemonitoring for frail patients with chronic diseases

SUMMARY:
The purpose of this study is to evaluate whether telemonitoring of frail patients with chronic diseases produces benefits in terms of reduced readmissions, improved health related quality of life, and improved health status. In addition, the trial evaluates the economic and organisational impact of the telemonitoring service and examines its acceptability by patients and health professionals.

DETAILED DESCRIPTION:
The study is designed to evaluate the impact of telemonitoring on the follow-up of elderly patients with one or more chronic diseases among heart failure, chronic obstructive pulmonary disease and diabetes. The particular target of patients selected has the particularity of being "frail" according to a set of social eligibility criteria, agreed by the clinicians participating at the study. General practitioners are the first clinicians in charge of managing these patients during the trial follow-up. The term of comparison is represented by a control group, followed by outpatient usual care.

From a clinical point of view, the trial will investigate how the remote monitoring of some clinical parameters contributes to reduce the access to healthcare facilities (emergency and planned hospitalization, bed-days, ER, specialist and GP visits), to improve the patients health-related quality of life and to reduce the anxiety about health conditions. A cost-effectiveness and cost-utility analysis will be carried out in order to determine if and how telemonitoring helps to limit the healthcare expenditure. The evaluation will deal also with organizational changes and task shift due to telemonitoring introduction and patients and professionals perception towards the service.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Diagnosis of one or more of the following chronic diseases:

  * Heart failure - diagnosis confirmed by echocardiogram or by a specialist assessment
  * Type 1 or 2 diabetes - with HbA1C of 7.5 or greater in the previous 15 months
  * Chronic Obstructive Pulmonary Disease (COPD) - diagnosis confirmed by spirometry and FEV1 ≤ 70% of predicted normal and/or FEV1/FVC ratio ≤ 70% or by a specialist assessment
* and at least one of the following Social inclusion criteria:

  * Have had a fall in the previous year or who are considered at high risk of falling
  * Need home social care
  * Have a caregiver who have difficulties to take care of him/her properly
  * Cognitive impairment/confusion, but with caregiver able to use devices.

Exclusion Criteria:

* Patient unable to use the telemonitoring equipment (alone and assisted)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 152 (Actual)
Dates: Start 2012-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Number of emergency hospitalisations | 12 months

SECONDARY OUTCOMES:
Number of primary care visits. | 12 months
Health related quality of life as measured by the SF 36 version 2 questionnaire | 12 months
All cause mortality | 12 months
Number of visits to emergency department | 12 months
Number of elective hospital admissions | 12 months
Number of bed days for hospitalised patients | 12 months
Anxiety and depression status as measured by Hospital Anxiety and Depression Scale, HADS. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicolò Seminara, MD, Principal Investigator — SIMG - LHA 9 of Treviso
Locations (7):
- Italy (7):
  - Local Heath Authority of Padova, Padua, Padova
  - Local Health Authority of Pieve di Soligo, Pieve di Soligo, Treviso
  - Local Health Authority of Treviso, Treviso, Treviso
  - Local Health Authority of Mirano, Mirano, Venezia
  - Local Heath Authority Veneziana, Venezia, Venezia
  - Local Heath Authority of Verona, Verona, Verona
  - Local Heath Authority of Thiene, Thiene, Vicenza